CLINICAL TRIAL: NCT00687817
Title: A Phase II Safety and Efficacy Study of Bavituximab Plus Paclitaxel and Carboplatin in Patients With Previously Untreated Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Bavituximab Plus Paclitaxel and Carboplatin in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: A.J. Leyco, RN/Associate Director, Clinical Affairs, Peregrine Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 0701
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — bavituximab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bavituximab plus paclitaxel and carboplatin — Weekly bavituximab dose of 3 mg/kg until disease progression, and up to 6 cycles of carboplatin at a dose of AUC=5 and paclitaxel 175 mg/m2 every 21 days (21-day cycles)

SUMMARY:
The primary objective of this study is to determine the overall response rate (complete response + partial response) to a combination of bavituximab plus carboplatin and paclitaxel in patients with previously untreated locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults over age 18 years of age with a life expectancy of at least 3 months
* Histologically or cytologically confirmed non-small cell lung cancer at stage IIIB (with pleural effusion), stage IV, or recurrence
* Measurable disease on cross sectional imaging at least 2 cm in longest diameter (1 cm if measured by spiral CT)
* Adequate hematologic (ANC ≥ 1500 cells/µL; Hemoglobin ≥9 g/dL; platelets ≥100,000/µL and ≤500,000/µL ), renal (serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 60 mL/min), and hepatic function (bilirubin ≤ 1.5 x ULN, ALT ≤ 3 x ULN, AST ≤ 3 x ULN)
* D-dimer ≤ 2 x ULN

Key Exclusion Criteria:

* Small cell or mixed histology
* Known history of bleeding diathesis or coagulopathy
* Any current evidence of clinically significant bleeding defined as gross hematuria, hemoptysis, or GI bleeding
* Any history of thromboembolic events (e.g., deep vein thrombosis or pulmonary thromboembolism)
* Prior chemotherapy, immunotherapy or radiotherapy to an area of measurable disease unless disease had recurred after radiotherapy
* Radiotherapy within 2 weeks preceding Study Day 1
* Symptomatic or clinically active CNS disease or metastatic lesions
* Major surgery within 4 weeks of Study Day 1
* Uncontrolled intercurrent disease (e.g., diabetes, hypertension, thyroid disease)
* Any history of angina pectoris, coronary artery disease or cerebrovascular accident, or transient ischemic attack
* A history of any condition requiring anti-platelet therapy with the exception of general cardiovascular prophylaxis with aspirin. Anti-platelet agents are prohibited during the study.
* Requirement for chronic daily treatment with NSAIDs, anti-platelet drugs, or steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Overall response (complete response + partial response) to a combination of bavituximab plus carboplatin and paclitaxel in patients with previously untreated locally advanced or metastatic non-small-cell lung cancer | one year

SECONDARY OUTCOMES:
Time to tumor progression, duration of response, overall survival and safety | Approximately 1 year

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - Apollo Hospital, Bannerghatta Rd, Banglore
  - Kidwai Hospital, Munigowda Road, Banglore
  - M S Ramaiah Hospital, New BEL Rd, Banglore
  - Bangalore Institute of Oncology Speciality Centre, Sampangi Ram Nagar, Banglore
  - Nizam's Institute of Medical Sciences, Panjagutta, Hyderabad
  - Yashoda Hospital, Somājigūda, Hyderabad
  - RCC Medical College, Trivandrum, Kerala
  - Orchid Nursing Home, Phoolanbhaghan, Kolkata
  - Ruby Hall Clinic, Pune, Pune

REFERENCES:
- [Derived] Digumarti R, Bapsy PP, Suresh AV, Bhattacharyya GS, Dasappa L, Shan JS, Gerber DE. Bavituximab plus paclitaxel and carboplatin for the treatment of advanced non-small-cell lung cancer. Lung Cancer. 2014 Nov;86(2):231-6. doi: 10.1016/j.lungcan.2014.08.010. Epub 2014 Aug 24. PMID 25236982